CLINICAL TRIAL: NCT01954030
Title: A Phase 1/2 Trial of Carboxyamidotriazole Orotate (CTO) Alone or in Combination With Bevacizumab for Adult Patients With Recurrent Malignant Glioma Post-Bevacizumab Failure
Brief Title: Phase 1/2 CTO + Bevacizumab for Recurrent Glioma Post-Bevacizumab Failure
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated early due to funding reasons prior to completing Phase 1
Sponsor: Annick Desjardins (Other)
Collaborators: Tactical Therapeutics, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Annick Desjardins, Associate Professor, Duke University
Organization: Duke University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00044274
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Malignant Glioma (WHO Grade III or IV)
Keywords: Carboxyamidotriazole Orotate; CTO; Bevacizumab; Avastin; Malignant Glioma; Pro00044274; Desjardins; Duke; The Preston Robert Tisch Brain Tumor Center
MeSH Terms: conditions — Glioma; Lymphoma, Follicular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CTO and Bevacizumab (Phase 1) (Experimental): The combination of CTO with the standard dosing of bevacizumab of 10 mg/kg every 2 weeks among patients with recurrent malignant glioma (World Health Organization (WHO) grade III or IV) that have previously failed bevacizumab
  Interventions: Drug: CTO and Bevacizumab
- Phase 2: CTO alone (Phase 2) (Experimental): The first 25 patients will be treated with CTO alone at the maximum tolerated dose (MTD) established in the Phase 1 portion of the study.
  Interventions: Drug: CTO alone
- CTO and Bevacizumab (Phase 2) (Experimental): The second group of 25 patients will be treated with the combination of CTO at the MTD established in the Phase 1 portion of this study and standard dosing of bevacizumab.
  Interventions: Drug: CTO and Bevacizumab

INTERVENTIONS:
Drug: CTO and Bevacizumab
  Other Names: CTO; Carboxyamidotriazole Orotate; Bevacizumab; Avastin
  Arms: CTO and Bevacizumab (Phase 1); CTO and Bevacizumab (Phase 2)
Drug: CTO alone
  Other Names: CTO; Carboxyamidotriazole Orotate
  Arms: Phase 2: CTO alone (Phase 2)

SUMMARY:
The primary objectives of the study are to determine the maximum tolerated dose (MTD) of Carboxyamidotriazole Orotate (CTO) when combined with standard dosing of bevacizumab among patients with recurrent malignant glioma (WHO grade III or IV) that have previously failed bevacizumab (Phase 1); to determine the activity of CTO alone in bevacizumab-failure WHO grade IV malignant glioma patients (Phase 2, Arm 1); to determine the activity of CTO plus bevacizumab in bevacizumab-failure WHO grade IV malignant glioma patients (Phase 2, Arm 2).

This study was terminated early due to funding issues. At the time of termination, the study was still in Phase 1 and no MTD for the combination of CTO and bevacizumab had been determined for this population. Phase 2 will not proceed.

DETAILED DESCRIPTION:
In Phase 1 of the study, we will conduct a dose-escalation study of the combination of CTO with the standard dosing of bevacizumab among patients with recurrent malignant glioma (WHO Grade III or IV) that have previously failed bevacizumab. All patients will have also received standard treatment with radiation therapy and temozolomide prior to enrollment on study.

The Phase 2 portion of this study will investigate two novel treatment regimens sequentially. Each regimen will include 25 patients with recurrent WHO grade IV malignant glioma who have been treated in the past with standard radiation therapy, temozolomide, and bevacizumab. All patients must have failed therapy while on bevacizumab. Subjects in the first treatment regimen will receive CTO alone and subjects in the second treatment regimen will receive the combination of CTO and bevacizumab together.

Note: This study was terminated early due to funding issues. At the time of termination, the study was still in Phase 1 and no MTD for the combination of CTO and bevacizumab had been determined for this population. Phase 2 will not proceed.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 portion: Patients must have recurrent histologically confirmed diagnosis of World Health Organization (WHO) grade III or IV malignant glioma with no more than 3 prior progressions
* Phase 2 portion: Patients must have recurrent histologically confirmed diagnosis of WHO grade IV malignant glioma (glioblastoma or gliosarcoma) with no more than 3 prior progressions.
* Must have had a least 1 prior progression on a bevacizumab-containing regimen
* Age greater than or equal to 18 years
* Karnofsky ≥ 70%
* Bi-dimensionally measurable disease, as assessed by magnetic resonance imaging based on The Revised Assessment in Neuro-Oncology (RANO) criteria
* Absolute neutrophil count (ANC) ≥1000 cells/µl, Platelets ≥ 100,000 cells/µl (without transfusion within 14 days before enrollment)
* Adequate renal function as indicated by the following: Serum creatinine < 1.25 times upper limit of normal (ULN) or calculated creatinine clearance ≥ 50 ml/min; Urine dipstick for proteinuria < 2+ unless a 24-hour urine protein <1 g of protein is demonstrated
* Prothrombin time (PT) ≤ 1.5 x ULN and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN within 14 days prior to first study treatment for patients not receiving anti-coagulation. The use of full-dose oral or parenteral anticoagulants is permitted as long as the PT or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the first study treatment.
* For patients on corticosteroids, they must be on a stable dose for 7 days prior to anticipated start of study drug, and the dose should not be escalated over entry dose level, if clinically possible
* Signed informed consent approved by the Institutional Review Board
* No evidence of > grade 1 active central nervous system (CNS) hemorrhage on the baseline magnetic resonance imaging (MRI) or computed tomography (CT) scan
* Female patients must not be pregnant or breast-feeding. Female patients of childbearing potential (defined as < 2 years after last menstruation or not surgically sterile) must use a highly effective contraceptive method (allowed methods of birth control, [i.e. with a failure rate of < 1% per year] are implants, injectables, combined oral contraceptives, intra-uterine device (IUD) (only hormonal), sexual abstinence or vasectomized partner) during the trial and for a period of > 6 months following the last administration of trial drug(s). Female patients with an intact uterus (unless amenorrhea for the last 24 months) must have a negative serum pregnancy test within 48 hours prior to first study treatment.
* Fertile male patients must agree to use a highly effective contraceptive method (allowed methods of birth control [i.e. with a failure rate of < 1% per year] include a female partner using implants, injectables, combined oral contraceptives, IUDs [only hormonal], sexual abstinence or prior vasectomy) during the trial and for a period of > 6 months following the last administration of trial drugs.

Exclusion Criteria:

* Pregnancy or breast-feeding
* Co-medication that may interfere with study results, for example, immuno-suppressive agents other than corticosteroids
* Active infection requiring intravenous (IV) antibiotics within 7 days before enrollment
* Prior, unrelated malignancy requiring current active treatment with the exception of cervical carcinoma in situ and adequately treated basal cell or squamous cell carcinoma of the skin
* Taking cytochrome P450 3A4 (CYP3A4) inducers and moderate or strong inhibitors (Note: Corticosteroids are allowed, as long as patients have been on a stable dose for 7 days prior to anticipated start of study drug, and the dose should not be escalated over entry dose level, if clinically possible)
* Less than 12 weeks from radiation therapy, unless progressive disease outside of the radiation field or progression on 2 consecutive scans or histopathologic confirmation
* Treated with immunotherapeutic agents or vaccines within 4 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy
* Treated with alkylating agents within 4 weeks before enrollment or treated with daily or metronomic chemotherapy within 1 week before enrollment, unless the patient has recovered from the expected toxic effects of such therapy
* Prior chemotherapy (non-alkylating agents) within 2 weeks before enrollment, unless the patient has recovered from the expected toxic effects of such therapy
* Current, recent (within 4 weeks of the first infusion of this study) use of an experimental drug, unless the patient has recovered from the expected toxic effects of study therapy

Vascular endothelial growth factor (VEGF) Inhibitor-Specific Exclusion Criteria are:

* Inadequately controlled hypertension (defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 100 mmHg) within 28 days of first study treatment
* Prior history of hypertensive crisis, hypertensive encephalopathy, reverse posterior leukoencephalopathy syndrome (RPLS)
* Prior history of gastrointestinal perforation or abscess
* Clinically significant (active) cardiovascular disease, for example cerebrovascular accidents ≤ 6 months prior to study enrollment, myocardial infarction ≤ 6 months prior to study enrollment, unstable angina, New York Heart Association (NYHA) Grade 2 or greater congestive heart failure (CHF), or serious cardiac arrhythmia uncontrolled by medication or potentially interfering with protocol treatment
* History or evidence upon physical/neurological examination of central nervous system disease (for example, seizures) unrelated to cancer unless adequately controlled by medication or potentially interfering with protocol treatment
* Significant vascular disease (for example, aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to start of study treatment
* History of pulmonary hemorrhage/hemoptysis ≥ grade 2 (defined as ≥ 2.5 mL bright red blood per episode) within 1 month of first study treatment
* History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (in the absence of therapeutic anticoagulation)
* Current or recent (within 10 days of study enrollment) use of aspirin (> 325 mg/day), clopidogrel (> 75 mg/day) or equivalent. Prophylactic or therapeutic low molecular weight heparin (LMWH) is allowed.
* Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to first study treatment, or anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedure, for example, stereotactic biopsy, within 7 days of first study treatment; placement of a vascular access device, within 2 days of first study treatment
* History of intracranial abscess within 6 months prior to first study treatment
* History of active gastrointestinal bleeding within 6 months prior to first study treatment
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* Known hypersensitivity to any component of bevacizumab or CTO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Phase 1: Determine the Maximum Tolerated Dose (MTD) of CTO when combined with standard dosing of bevacizumab | 1 year
  A standard "3+3" design to determine the MTD of CTO in combination with bevacizumab. Subjects will be administered CTO orally on a continuous daily dosing schedule, while subjects will receive bevacizumab (10 mg/kg) every 2 weeks. Cohorts of 3-6 subjects will accrue at each dose level of CTO, beginning with 225 mg/m2, until MTD is defined. The MTD is the highest dose level at which ≤ 1 out of 6 experienced a dose limiting toxicity (DLT).
Phase 2: Percentage of subjects who remain alive and progression-free at 6 months | 2 years
  Percentage of participants surviving six months from start of study treatment without progression of disease. Progression-free survival (PFS) was defined as the time from start of study treatment to the date of the first documented progression according to the Response Assessment in Neuro-Oncology (RANO) criteria, or to death due to any cause.

SECONDARY OUTCOMES:
Phase 1: Number of subjects who experience a dose-limiting toxicity (DLT) during cycle 1 | 1 year
  All toxicities will be collected using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. DLTs will be defined as any of the following events that are possibly, probably, or definitely attributable to CTO or lomustine:
  Non-hematologic:
  * Nausea/vomiting of Grade 3 or greater despite maximal antiemetic therapy
  * Diarrhea of Grade 3 or greater despite maximal antidiarrheal therapy
  * Any other Grade 3 or 4 non-hematologic toxicity
  Hematologic:
  * Any Grade 4 neutropenia
  * Grade 3 neutropenia associated with fever of any duration or where significant sepsis results
  * Grade 4 thrombocytopenia
Phase 2: Percentage of subjects who experience a dose-limiting toxicity (DLT) during any cycle of protocol treatment | 2 years
  All toxicities will be collected using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. DLTs will be defined as any of the following events that are possibly, probably, or definitely attributable to CTO or lomustine:
  Non-hematologic:
  * Nausea/vomiting of Grade 3 or greater despite maximal antiemetic therapy
  * Diarrhea of Grade 3 or greater despite maximal antidiarrheal therapy
  * Any other Grade 3 or 4 non-hematologic toxicity
  Hematologic:
  * Any Grade 4 neutropenia
  * Grade 3 neutropenia associated with fever of any duration or where significant sepsis results
  * Grade 4 thrombocytopenia
Phase 2: Median Overall Survival (OS) | 2 years
  Time in months from start of study treatment to date of death due to any cause. Patients alive as of the last follow-up will have OS censored at the last follow-up date. Median OS will be estimated using a Kaplan-Meier curve.
Phase 2: 6 and 12 month Overall Survival (OS) | 2 years
  Percentage of participants surviving 6 and 12 months from start of study treatment. OS is defined as time from start of study treatment to the date of death due to any cause.
Phase 2: Percentage of subjects with best overall response (BOR) of complete response (CR) or partial response (PR) | 2 years
  Response is based on Response Assessment in Neuro-Oncology (RANO) criteria as determined by investigator assessment. A confirmation of response was not required. Complete Response was defined as complete disappearance on MR/CT of all enhancing tumor and mass effect, off all corticosteroids (or receiving only adrenal replacement doses), accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks. Partial Response was defined as greater than or equal to 50% reduction in tumor size on MR/CT by bi-dimensional measurement, on a stable or decreasing dose of corticosteroids, accompanied by a stable or improving neurologic examination, and maintained for at least 4 weeks.
Phase 2: Median PFS | 2 years
  Time in months from start of study treatment to the date of first progression according to RANO criteria, or to death due to any cause. Patients alive who had not progressed as of the last follow-up will have PFS censored at the last follow-up date. Median PFS will be estimated using a Kaplan-Meier curve.
Phase 2: 12 month PFS | 2 years
  Percentage of participants surviving six months from the start of study treatment without progression of disease. PFS is defined as the time from the date of study treatment initiation to the date of the first documented progression according to the RANO criteria, or to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke University
Locations (1):
- The Preston Robert Tisch Brain Tumor Center at Duke, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at Duke — http://www.cancer.duke.edu/btc/